CLINICAL TRIAL: NCT05543187
Title: An Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-625 in the Treatment of Subjects With Progressive Familial Intrahepatic Cholestasis
Brief Title: A Study of TAK-625 for the Treatment of Progressive Familial Intrahepatic Cholestasis (PFIC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-625-3002; jRCT2031220356 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Progressive Familial Intrahepatic Cholestasis (PFIC)
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAK-625, Primary cohort (Experimental): TAK-625 orally, twice daily (BID) for 4 weeks as Dose Escalation Period. The dose in Dose Escalation Period will be increased weekly, 150 mcg/kilograms (kg), 300 mcg/kg, 450 mcg/kg, and 600 mcg/kg. After Dose Escalation Period, TAK-625 600 mcg/kg (or maximum tolerated dose [MTD]), orally, BID up to study completion.
  Interventions: Drug: TAK-625
- TAK-625, Supplemental cohort (Experimental): TAK-625 orally, twice daily (BID) for 4 weeks as Dose Escalation Period. The dose in Dose Escalation Period will be increased weekly, 150 mcg/kilograms (kg), 300 mcg/kg, 450 mcg/kg, and 600 mcg/kg. After Dose Escalation Period, TAK-625 600 mcg/kg (or maximum tolerated dose [MTD]), orally, BID up to study completion.
  Interventions: Drug: TAK-625

INTERVENTIONS:
Drug: TAK-625 — TAK-625 orally, twice daily (BID)
  Other Names: Maralixibat chloride

SUMMARY:
The main aim of the study is to check if TAK-625 improves symptoms of Progressive Familial Intrahepatic Cholestasis (PFIC), side effect from the study treatment or TAK-625, and how much TAK-625 stays in their blood over time. This will help the study sponsor (Takeda) to work out the best dose to give people in the future.

The participants will be treated with TAK-625 for up to the end of study (about 34 months).

Participants will visit their study clinic 15 times from the start of study. After 15 times visits, participants will visit their study clinic every 12 weeks up to the end of study.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is Japanese male or female with a body weight >=3.0 kg and who is >=1 month of age at the time of informed consent.
2. The participant has a cholestasis as manifested by total serum bile acid (sBA) >=3^ upper limit of the normal range (ULN) (applies to the primary cohort only).
3. The participant has an average morning ItchRO (Obs) score >=1.5 during 4 consecutive weeks of the screening period, leading to the baseline visit (Week 0/Visit 2). Since it is difficult to evaluate pruritus in infants, participants <12 months of age at screening whose pruritus is unavoidably difficult to be evaluated are not necessarily required to meet the above score.
4. The caregiver has completed at least 21 valid* morning ItchRO (Obs) entries during 4 consecutive weeks of the screening period, leading to the baseline visit (Week 0/Visit 2) (*valid=completed and not answered as "I don't know"; the maximum allowed invalidreports=7, no more than 2 invalid reports during the last 7 days before the baseline visit [Week 0/Visit 2]).
5. The participant has a diagnosis of progressive familial intrahepatic cholestasis (PFIC) based on:

   Chronic cholestasis as manifested by persistent (>6 months*) pruritus in addition to biochemical abnormalities and/or pathological evidence of progressive liver disease. (* =<6 months is acceptable for participants <12 months of age).

   AND

   For Primary cohort:

   a) The participant has a genetic testing result consistent with disease-causing variation in ABCB11 (PFIC2), based on a genotyping.

   For Supplemental cohort:
   1. The participant has a genetic testing results consistent with disease causing variation in ATP8B1 (PFIC1), ABCB4 (PFIC3), or tight junction protein 2 gene (TJP2) (PFIC4), based on a genotyping.
   2. The participant has a PFIC phenotype without a known mutation or with another known mutation not described above.
   3. The PFIC participant has internal or external biliary diversion surgery history, and the internal or external biliary diversion surgery was reversed.
6. The participant (whenever possible) and caregiver are able to be contacted by phone for scheduled remote visits (participant contacts [phone calls]).
7. Both a caregiver and participant above the age of assent are capable of reading and understanding the questionnaires.
8. The same caregiver should be contacted during this study. The ItchRO (Obs) should be completed by the same caregiver for consistency during this study, even if the participant is an adult (over 18 years old).

Exclusion Criteria:

1. The diagnosed with PFIC2 due to ABCB11 mutation that predicts complete absence of BSEP function due to the type of ABCB11 mutation (t-PFIC2), based on a genotyping (applies to the primary cohort only).
2. The participant has a diagnosis of benign recurrent intrahepatic cholestasis indicated by a history of intermittent cholestasis with no disease progression.
3. The participant has a current or recent history (<1 year) of atopic dermatitis or other non-cholestatic diseases associated with pruritus.
4. The participant has a previous history of surgical interruption of the enterohepatic circulation (applies to the primary cohort only).
5. The participant with chronic diarrhea requiring intravenous (IV) fluid or nutritional intervention and/or its sequelae at screening or during the 6 months prior to screening.
6. The participant has a history of liver transplant or currently requires imminent liver transplant.
7. The participant with decompensated cirrhosis (international normalized ratio [INR] >1.5, and/or albumin <30 g/L, history, or presence of clinically significant ascites, and/or variceal hemorrhage, and/or encephalopathy).
8. The participant has an alanine aminotransferase (ALT) or total serum bilirubin (TSB) level >15^ ULN at screening.
9. The participant has other liver disease.
10. The participant has any other disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, including bile salt metabolism in the intestine (eg, inflammatory bowel disease), per investigator discretion.
11. The participant has a possible malignant liver mass in imaging, including screening ultrasound.
12. The participant has received bile acid, lipid binding resins or ileal bile acid transporter (IBAT) inhibitors within 28 days prior to screening and throughout the trial.
13. The participant who has received sodium phenylbutyrate for less than 6 months at the initiation of screening.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2025-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- Japan (8):
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Tsuyama Chuo Hospital, Tsuyama, Okayama-ken
  - Osaka University Hospital, Suita, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Kyoto University Hospital, Kyoto
  - Saitama Prefectural Children's Medical Center, Saitama

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5c64837a6d7c464c

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 sites in Japan from 10 January 2023 to 22 July 2025.
Pre-assignment Details: Participants diagnosed with progressive familial intrahepatic cholestasis 2 (PFIC2) due to adenosine triphosphate (ATP) binding cassette subfamily B member 11 (ABCB11) mutation that predicted residual bile salt excretion pump (BSEP) function (non-truncating [nt]-PFIC2) were enrolled in Primary Cohort, and participants with other PFIC subtypes or post-surgical were enrolled in Supplemental Cohort, to receive TAK-625 twice daily (BID).
Groups:
- Primary Cohort: TAK-625: Participants diagnosed with PFIC2 due to ABCB11 mutation that predicted residual BSEP function received TAK-625 orally, BID. In dose escalation period, dose was increased weekly, 150 micrograms per kilograms (mcg/kg), 300 mcg/kg, 450 mcg/kg, and 600 mcg/kg for up to 4 weeks (Weeks 1 to 4) or extended to 6 weeks depending on the safety or tolerability concerns. After the dose escalation period, each participant continued dosing with TAK-625 600 mcg/kg, orally, BID dose level in the stable dosing period, a follow-up dosing period after Week 48, and a safety follow-up period.
- Supplemental Cohort: TAK-625: Participants diagnosed with other PFIC subtypes or post-surgical received TAK-625 orally, BID. In dose escalation period, dose was increased weekly, 150 mcg/kg, 300 mcg/kg, 450 mcg/kg, and 600 mcg/kg for up to 4 weeks (Weeks 1 to 4) or extended to 6 weeks depending on the safety or tolerability concerns. After the dose escalation period, each participant continued dosing with TAK-625 600 mcg/kg, orally, BID dose level in the stable dosing period, a follow-up dosing period after Week 48, and a safety follow-up period.
Period: Overall Study
Arm/Group | Primary Cohort: TAK-625 | Supplemental Cohort: TAK-625
Started | 3 | 2
Dosed TAK-625 150 mcg/kg (TAK-625 orally, BID for 1 week in Dose Escalation Period.) | 3 | 2
Dosed TAK-625 300 mcg/kg (TAK-625 orally, BID for 1 week in Dose Escalation Period.) | 3 | 2
Dosed TAK-625 450 mcg/kg (TAK-625 orally, BID for 1 week in Dose Escalation Period.) | 3 | 2
Dosed TAK-625 600 mcg/kg (TAK-625 orally, BID for 1 week in Dose Escalation Period and for up to 22 weeks after Dose Escalation Period.) | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) included all participants who received at least one dose of study drug. As per-planned analysis, the cohort-wise (primary and supplemental) data were analyzed, collected, and reported in this study.
Groups:
- Primary Cohort: TAK-625: Participants diagnosed with PFIC2 due to ABCB11 mutation that predicted residual BSEP function received TAK-625 orally, BID. In dose escalation period, dose was increased weekly, 150 mcg/kg, 300 mcg/kg, 450 mcg/kg, and 600 mcg/kg for up to 4 weeks (Weeks 1 to 4) or extended to 6 weeks depending on the safety or tolerability concerns. After the dose escalation period, each participant continued dosing with TAK-625 600 mcg/kg, orally, BID dose level in the stable dosing period, a follow-up dosing period after Week 48, and a safety follow-up period.
- Total: Total of all reporting groups
Arm/Group | Primary Cohort: TAK-625 | Supplemental Cohort: TAK-625 | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (3.21) | 8.0 (4.24) | 7.8 (3.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in the Average Morning Itch Reported Outcome (ItchRO) (Observer Instrument [Obs]) Severity Score Between Baseline and the Average of Week 15 Through Week 26
Description: The ItchRO (Obs) scale measures severity of pruritus. The score on ItchRO (Obs) scale ranged from 0 to 4, where 0=None observed or reported, 1=Mild, 2=Moderate, 3=Severe, 4=Very severe. A higher score indicated more severe pruritus. Average baseline morning ItchRO (Obs) scores were calculated as sum of the morning scores divided by number of morning scores for the 4-week (28 days) time periods (that is [i.e.], Day -28 to Day -1). Average morning ItchRO (Obs) scores Week 15 through Week 26 were calculated as the sum of the morning scores divided by the number of morning scores from Week 15 to Week 26. Change was calculated as: Average value of Weeks 15 to 26 - Average value of Baseline (Day -28 to Day -1).
Time Frame: Baseline to Week 15 through Week 26
Population: ITT included all participants who received at least one dose of study drug. As per-planned analysis, the cohort-wise (primary and supplemental) data were analyzed, collected, and reported in this study.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Cohort: TAK-625 | Supplemental Cohort: TAK-625
Number analyzed (Participants) | 3 | 2
score on a scale | -1.514 [-3.6541 to 0.6255] | -0.202 [-3.6957 to 3.2911]

2. Secondary Outcome: Change in the Average Morning ItchRO (Obs) Frequency Score Between Baseline and the Average of Week 15 Through Week 26
Description: The ItchRO (Obs) scale measures frequency of pruritus. The score on ItchRO (Obs) scale ranged from 0 to 4, where 0=None observed or reported, 1= A little bit of the time, 2= Some of the time, 3= Most of the time, 4= Almost all of the time/constantly, I don't know) to describe their pruritus condition. 'I don't know' was categorized as missing data. A higher score indicated more severe pruritus. Baseline average morning ItchRO (Obs) frequency scores were calculated as the sum of the morning frequency scores divided by the number of morning severity scores for the 4-week (28 days) time periods. (i.e., Day -28 to Day -1). Average morning ItchRO (Obs) frequency scores of Week 15 through Week 26 were calculated as the sum of the morning frequency scores divided by the number of mornings frequency scores from Week 15 to Week 26. Change was calculated as: Average value of Weeks 15 to 26 - Average value of Baseline (Day -28 to Day -1).
Time Frame: Baseline to Week 15 through Week 26
Population: ITT included all participants who received at least one dose of study drug. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. As per-planned analysis, the cohort-wise (primary and supplemental) data were analyzed, collected, and reported in this study.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Cohort: TAK-625 | Supplemental Cohort: TAK-625
Number analyzed (Participants) | 2 | 2
score on a scale | -0.740 [-4.8063 to 3.3254] | -0.735 [-6.0922 to 4.6213]

3. Secondary Outcome: Change From Baseline in Total Serum Bile Acid (sBA) Levels to Week 26
Description: Change from baseline was calculated as: Post-baseline observed value - Baseline (before first dosing) observed value. Change from baseline in total sBA levels to Week 26 was reported.
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: micromoles per liter (mcmol/L)
Arm/Group | Primary Cohort: TAK-625 | Supplemental Cohort: TAK-625
Number analyzed (Participants) | 3 | 2
micromoles per liter (mcmol/L) | -149.900 [-561.4008 to 261.6008] | -18.250 [-173.9010 to 137.4010]

4. Secondary Outcome: Percentage of Participants (Responders) Who Experienced an sBA Control From Baseline Through Week 26
Description: Responders to sBA control were defined as participants who achieved a decrease to less than (<) 102 mcmol/L, a decrease of greater than (>) 75 percentage (%), or normalization at any timepoint from baseline through Week 26.
Time Frame: Baseline through Week 26
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Cohort: TAK-625 | Supplemental Cohort: TAK-625
Number analyzed (Participants) | 3 | 2
percentage of participants | 33.3 [0.84 to 90.57] | 0.0 [0.00 to 84.19]

5. Secondary Outcome: Change in the ItchRO (Obs) Weekly Average Severity Between Baseline and the Average of Week 15 Through Week 26
Description: ItchRO (Obs) scale measures severity of pruritus, score ranged from 0 to 4, where 0=None observed or reported, 1=Mild, 2=Moderate, 3=Severe, 4=Very severe. A higher score indicated more severe pruritus. Weekly average severity was calculated based on daily maximum severity scores from both morning and evening. Average baseline morning and evening ItchRO (Obs) scores were calculated as sum of morning or evening scores divided by number of morning or evening scores for 4-week (28 days) time periods (i.e., Day -28 to Day -1). Average morning and evening ItchRO (Obs) scores Week 15 to Week 26 were calculated as sum of morning or evening scores divided by number of morning or evening scores from Week 15 to Week 26. Change was calculated as: Average value of Weeks 15 to 26 - Average value of Baseline (Day -28 to Day -1).
Time Frame: Baseline to Week 15 through Week 26
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Cohort: TAK-625 | Supplemental Cohort: TAK-625
Number analyzed (Participants) | 3 | 2
score on a scale | -1.629 [-3.5064 to 0.2481] | -0.254 [-4.3906 to 3.8824]

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (up to Week 133)
Description: As per-planned analysis, the cohort-wise (primary and supplemental) data were analyzed, collected, and reported in this study.
Arm/Group | Primary Cohort: TAK-625 | Supplemental Cohort: TAK-625
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Cohort: TAK-625 (N=3) | Supplemental Cohort: TAK-625 (N=2)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Auricular haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Otitis media (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Viral pharyngitis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT05543187/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT05543187/SAP_002.pdf